CLINICAL TRIAL: NCT04980638
Title: A Prospective, Open-label, Genotype-match Controlled, Multicenter Clinical Trial to Investigate the Efficacy and Safety of Intra-amniotic ER004 as a Prenatal Treatment for Male Subjects With XLHED
Brief Title: Intraamniotic Administrations of ER004 to Male Subjects With X-linked Hypohidrotic Ectodermal Dysplasia
Acronym: EDELIFE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: EspeRare Foundation (Other)
Collaborators: Pierre Fabre Medicament (Industry); Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ER004-CLIN01/F60082AI201
Record Dates: First submitted 2021-07-20; First posted 2021-07-28 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: X-Linked Hypohidrotic Ectodermal Dysplasia (XLHED)
MeSH Terms: conditions — Ectodermal Dysplasia 1, Anhidrotic

STUDY DESIGN:
Intervention Model Description: This is an open-label, single-arm, genotype-match controlled for primary estimand, non randomized study. The primary efficacy outcome will be compared to genotype matched untreated male relatives with XLHED or to genotype-matched controls from an external XLHED database (clinical and natural history studies from which untreated genotype-matched controls will be identified).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ER004 (Experimental): Human immunoglobulin G1 constant region - human ectodysplasin-A1 receptor binding domain fusion protein.
  Interventions: Biological: ER004

INTERVENTIONS:
Biological: ER004 — Intra-amniotic route 100 mg/kg of estimated fetal weight per injection. 3 injections, approximately 3 weeks apart starting from gestational week 26

SUMMARY:
This is an open-label, prospective, genotype-match controlled for primary estimand, non randomized, multicenter, international Phase 2 clinical trial designed to investigate the efficacy and safety of ER004 administered intraamniotically as a treatment for unborn XLHED male subjects.

DETAILED DESCRIPTION:
X-linked hypohidrotic ectodermal dysplasia (XLHED) is a rare developmental disease affecting body parts derived from the embryonal ectoderm. It is caused by a broad spectrum of mutations in the ectodysplasin A gene (EDA). The main symptoms of XLHED are hypo- or anhidrosis, oligo- or anodontia, and hypotrichosis. Current treatment options are limited to the management of disease symptoms and prevention of complications. Effective corrective treatment for XLHED remains a high unmet medical need. ER004 represents a first-in-class signaling protein replacement molecule designed for specific, high affinity binding to the endogenous EDA1 receptor (EDAR). The proposed mechanism of action of ER004 is the replacement of the missing EDA1 protein in patients with XLHED. The aim of this prospective, open-label, genotype-match controlled, multicenter Phase 2 trial is to confirm the efficacy and safety results for ER004 administered intra-amniotically in a larger cohort of subjects. The target population will consist of male XLHED fetuses/subjects with EDA mutation confirmed by genetic diagnosis of a mutation in one of the maternal EDA alleles and ultrasonographic diagnosis of a significantly reduced number of fetal tooth germs, or by documented direct genetic diagnosis of a hemizygous EDA mutation. In the main study phase, efficacy and safety of the treated subjects will be assessed up to 6 months of age and safety of the mothers will be assessed up to 1 month after delivery of the child. In long-term follow-up phase, efficacy and safety of the treated subjects will be assessed up to 5 years of age. Treated subjects sweating ability will be compared to an untreated relative from his family, when available, or from a matched controlled subject from a previous natural history.

ELIGIBILITY:
Inclusion Criteria:

For mother: adult mother with confirmed pregnancy no later than week 23+6 and genetically confirmed as carrier of an EDA mutation

* For fetal subject : male fetal subject with confirmed diagnosis of XLHED
* For untreated relative: untreated male relative subject aged between 6 months and 75 years with the same EDA mutation as the treated subject

Exclusion Criteria:

* For mother: any evidence of active maternal infection associated with a risk of preterm birth and/or congenital anomalies of prenatal and postnatal risk to the child. Documented maternal HIV infection. Any pre-existing maternal medical condition that increases the risk of preterm birth or increases the risk of a serious untoward event occurring to the mother during pregnancy. Any pregnancy disorder associated with an increased risk of preterm birth, and/or maternal, fetal or neonatal morbidity/mortality.
* For fetal subject : second major anatomic anomaly (not related to the underlying XLHED) that contributes to a significant morbidity or mortality risk, or echocardiogram or ultrasonography or other findings that indicate a high risk of fetal demise or risk of preterm birth. Any condition other than XLHED that is likely to have an impact on the number of tooth germs. Any other medical condition which in the opinion of the investigator would not allow for safe conduct of the study for the subject, or that would interfere with efficacy assessments.
* For untreated relative: carrier of an hypomorphic EDA mutation. Known hypersensitivity to pilocarpine or pilocarpine-like muscarinic agonists. Presence of an implanted device (e.g., defibrillator, neurostimulator, pacemaker). Previous treatment with the study intervention by any route of administration prior to study start.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant female
Enrollment: 20 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Mean sweat volume | at 6 months of age (corrected age for subjects born at < 37 weeks)
  For treated subject, mean sweat volume is collected on both forearms after local stimulation with pilocarpine (pilocarpine-induced sweating)

SECONDARY OUTCOMES:
Mean sweat pore density (number/cm2) | at 6 months of age (key secondary) and other timepoints : 3, 12, 18, 24, 36, 48 and 60 months of age (secondary)
  Mean sweat pore density (number/cm2) determined by direct visualization with a VivaScope® at 2 different sites on the sole/soles of the foot/feet (up to 12 months) or at 2 different sites on the sole/soles of the foot/feet and/or palm/palms of the hand/hands (>12 months)
Dental development | at 6 months of age (key secondary) and other timepoints : 12, 18, 24, 36, 48 and 60 months of age (secondary)
  Dental development evaluated by the number of erupted teeth and tooth germs (palpable alveolar structures in the alveolar ridge) as determined by dental examination
Mean sweat volume | At 3, 12, 18, 24, 36, 48, 60 months of age
  For treated subject, mean sweat volume is collected on both forearms after local stimulation with pilocarpine (pilocarpine-induced sweating)
Number of Meibomian glands | At 6 and 60 months of age
  Number of Meibomian glands in the lower eyelids determined by Meibography
Ocular surface assessment | At 24, 48 and 60 months of age
  Ocular surface assessment (normal, keratitis superficialis punctate) by eye using fluorescein
Tear film break-up time | At 24, 48 and 60 months of age
  Tear film break-up time (seconds) determined using fluorescein
Ocular Surface Disease Index (OSDI) score | At 60 months of age
  Score assessed on a scale of 0 to 100 through the OSDI questionnaire. Higher scores mean a worse outcome
Salivation | At 60 months of age
  Saliva (volume and flow rate) assessed with Quantisal oral fluid collection device
XLHED-related hospitalizations | Up to 60 months of age
  XLHED-related hospitalisation because of hyperthermia or because of unexplained fever, respiratory, skin, eye or ear infections
Assessment of eczema | At different timepoints from 6 to 60 months of age
  Eczema will be assessed using the EASI score
Incidence of TEAEs (treatment-emergent adverse events) | Up to 60 months of age
  Number of subjets with TEAEs
Incidence of TESAEs (treatment-emergent serious adverse events) | Up to 60 months of age
  Number of subjects with TESAEs
Incidence of TEAEs (treatment-emergent adverse events) leading to treatment discontinuation | Up to 60 months of age
  Number of subjects with TEAEs leading to treatment discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Holm Schneider, MD, Principal Investigator — University Erlangen-Nürnberg Erlangen, Germany
Locations (8):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Washington University, St Louis, Missouri
- Hôpital Necker - Enfants Malades, Paris, Paris, France
- Germany (2):
  - Universitaetsklinikum Erlangen, Erlangen, Bavaria
  - Universitaetsklinikum Leipzig AoeR, Leipzig, Saxony
- IRCCS Ca' Granda Ospedale Policlinico, Milan, Italy
- Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia, Spain
- University Hospital of Wales Cardiff and Vale University Local Health, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schneider H, Faschingbauer F, Schuepbach-Mallepell S, Korber I, Wohlfart S, Dick A, Wahlbuhl M, Kowalczyk-Quintas C, Vigolo M, Kirby N, Tannert C, Rompel O, Rascher W, Beckmann MW, Schneider P. Prenatal Correction of X-Linked Hypohidrotic Ectodermal Dysplasia. N Engl J Med. 2018 Apr 26;378(17):1604-1610. doi: 10.1056/NEJMoa1714322. PMID 29694819
- [Background] Schneider H, Hadj-Rabia S, Faschingbauer F, Bodemer C, Grange DK, Norton ME, Cavalli R, Tadini G, Stepan H, Clarke A, Guillen-Navarro E, Maier-Wohlfart S, Bouroubi A, Porte F. Protocol for the Phase 2 EDELIFE Trial Investigating the Efficacy and Safety of Intra-Amniotic ER004 Administration to Male Subjects with X-Linked Hypohidrotic Ectodermal Dysplasia. Genes (Basel). 2023 Jan 6;14(1):153. doi: 10.3390/genes14010153. PMID 36672894
- [Background] Schneider H, Schweikl C, Faschingbauer F, Hadj-Rabia S, Schneider P. A Causal Treatment for X-Linked Hypohidrotic Ectodermal Dysplasia: Long-Term Results of Short-Term Perinatal Ectodysplasin A1 Replacement. Int J Mol Sci. 2023 Apr 12;24(8):7155. doi: 10.3390/ijms24087155. PMID 37108325
- See also: EDELIFE Study website (Germany) — http://www.EDELIFEklinischestudie.com/
- See also: EDELIFE Study website (France) — http://www.essaicliniqueEDELIFE.com/
- See also: EDELIFE Study website (Spain) — http://www.ensayoclinicoEDELIFE.com/
- See also: EDELIFE Study website (UK) — http://www.EDELIFEclinicaltrial.com/
- See also: EDELIFE Study website (Italy) — http://www.studioclinicoEDELIFE.com
- See also: EDELIFE Study website (USA) — http://www.EDELIFEclinicaltrial.com/